CLINICAL TRIAL: NCT00359125
Title: Efficacy of Mifepristone (RU-486) in the Treatment of Bipolar Depression.
Brief Title: RU-486 in the Treatment of Bipolar Depression
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Western Economic Diversification Canada (Other Government); Stanley Medical Research Institute (Other)
Responsible Party: Dr. Allan Young, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C06-0327; H06-0093; NCT00363064 (obsolete NCT alias)
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Bipolar Depression
Keywords: bipolar; RU-486; mifepristone; neurocognition; mood; cortisol; HPA axis
MeSH Terms: conditions — Bipolar Disorder | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): RU-486, 600 mg/day for 1 week.
  Interventions: Drug: mifepristone (RU-486)
- 2 (Placebo Comparator): Placebo, 600 mg/day for 1 week
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: mifepristone (RU-486) — RU-486, 600 mg/day for 1 week.
  Other Names: Mifepristone
  Arms: 1
Other: Placebo — Placebo, 600 mg/day for 1 week.
  Arms: 2

SUMMARY:
Bipolar disorder is a chronic and recurrent illness which involves episodes of mania and depression. It is believed that disturbance of the stress hormone system (the hypothalamic-pituitary-adrenal or HPA axis) may cause thinking and memory problems and make the depressive symptoms worse in bipolar disorder. Early studies have shown that mifepristone may have antidepressant effects (may improve the symptoms of depression) and may also maintain or enhance cognition (memory and thinking functions).

The purpose of this study is to determine the potential therapeutic efficacy (usefulness) of mifepristone in bipolar depression by assessing the effects of the medication on depressive symptoms and on cognition. This will be done by questionnaires and thinking tests.

This study will also try to clarify the functional changes that accompany bipolar disorder by analyzing saliva samples (assessing the stress response by measuring the levels of 2 stress hormones: cortisol and DHEA).

DETAILED DESCRIPTION:
Detailed Description:

This study will be a parallel design randomized control trial. Duration of study is 10 weeks per subject. Following a baseline assessment of neurocognitive performance, mood symptoms, and neuroendocrine functioning (HPA axis functioning), bipolar depressed outpatients (n=100) will be randomized (week 0) to receive either mifepristone 600 mg daily (n=50) or matching placebo (n=50) for 7 days. Outcome measures will be completed at baseline (pre-medication), at the time of anticipated main response (week 3, i.e. 2 weeks after cessation of treatment), and at week 8 (to determine the persistence of any effects).

Neurocognitive performance (pre and post mifepristone treatment) will be evaluated with tests that have previously been shown to be affected by corticosteroids and to be abnormal in bipolar disorder. The neurocognitive battery will measure learning and memory, attention, executive functioning, and facial expression (which has been shown to be a sensitive measure of affective shift).

Mood symptoms will be evaluated at every study visit using standard clinician and patient self-rated scales.

Neuroendocrine functioning (HPA axis functioning) will be measured by the dexamethasone suppression test (DST) response to dexamethasone. This is a measure of the function of the glucocorticoid receptor. Subjects will also be asked for salivary samples to measure the cortisol response to wakening and the ratio of cortisol to the protective steroid DHEA. These validated tests will be used to improve our understanding of the mechanism of the therapeutic effect of mifepristone.

Fifty (50) matched-healthy controls will also undergo the baseline assessments of neurocognitive performance, mood symptoms, and neuroendocrine functioning. They will provide information about the pathophysiology of bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

Male & female outpatients between 19-65 years of age with a diagnosis of bipolar depression. Women must not be currently pregnant and must use a reliable method of contraception for the duration of the study. Subjects must be on stable medication (4 weeks minimum) for their bipolar illness. Subjects must be able to provide written informed consent. Subjects must adequately understand written & verbal English as rating scales as neurocognitive tests are only in English.

Exclusion Criteria:

Those not meeting the above criteria and those not competent to give informed consent. Women who are currently pregnant. Also excluded: those who have a clinically significant medical illness (including significant head injury with loss of consciousness), those at immediate risk of harming self or others, are currently abusing alcohol or drugs, those with a neurological disorder or uncompensated endocrine disorder, those with a known allergy to mifepristone, those currently being treated with an investigational medication or medication that is contraindicated with mifepristone.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive performance at weeks -1, 3 & 8 and symptom change at weeks -2, -1, 0, 1, 2, 3, 4, 5 & 8

SECONDARY OUTCOMES:
HPA axis functioning from saliva samples at weeks -2, -1, 2, 3 & 8

CONTACTS AND LOCATIONS:
Overall Officials: Allan Young, MD, Principal Investigator — The University of British Columbia
Locations (1):
- University of British Columbia, Dept. of Psychiatry, Vancouver, British Columbia, Canada